CLINICAL TRIAL: NCT02681133
Title: How is Physical Activity Level and Educational Expectations of Patient With Knee Osteoarthritis : Epidemiological Study in Spa Therapy
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Innovatherm (Industry)
Responsible Party: Sponsor
Other Study IDs: CHU-0256
Record Dates: First submitted 2016-02-05; First posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Knee Osteoarthritis; Physical Activity
Keywords: Physical activity level; Knee osteoarthritis; Non pharmacological treatment; Survey; Socio-demographic, clinical variables; Barriers, facilitators Fears and beliefs; Function
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- patients with knee pain
  Interventions: Other: Epidemiological study Survey

INTERVENTIONS:
Other: Epidemiological study Survey

SUMMARY:
The primary purpose is to evaluate the level of physical activity in patients with knee osteoarthritis in a spa treatment and doing epidemiological study about this patient.

DETAILED DESCRIPTION:
Explain the physical activity level of knee osteoarthritis by socio-demographic, clinical variables, barriers and facilitators of regular physical activity practice, fears and beliefs about their condition, functional limitations and physical inactivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, aged 50 to 75 years.
* Patients with knee pain reported to osteoarthritis
* Patient affiliated to a social security scheme (beneficiary entitled)
* Patient registered spa

Exclusion Criteria:

-

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with knee pain reported to osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Level of physical activity with IPAQ short form | During the spa treatment

SECONDARY OUTCOMES:
Socio-demographic variables as assessed by : age, sex, family situation, level of study | During the spa treatment
Fears and beliefs as assessed by KOFBeQ | During the spa treatment
Pain as assessed by EVA | During the spa treatment
Functional status as assessed by WOMAC | During the spa treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France